CLINICAL TRIAL: NCT00215176
Title: A Study of Modafinil for Atypical Depression
Brief Title: Modafinil for Atypical Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Cephalon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4428
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2005-09

CONDITIONS: Atypical Depression
Keywords: atypical depression; psychostimulants; modafinil
MeSH Terms: interventions — Modafinil

INTERVENTIONS:
Drug: modafinil

SUMMARY:
The purposes of the study are to: 1) evaluate the short-term efficacy and safety of modafinil in atypical depression; and 2) to evaluate the efficacy of modafinil in preventing relapse of atypical depression. The hypothesis is that modafinil is safe and effective in the treatment of atypical depression.

DETAILED DESCRIPTION:
This study on the safety and efficacy of modafinil on atypical depression has an initial 12-week open label treatment period with modafinil that is followed by a 12-week double-blind, randomized parallel treatment period with either modafinil or matching placebo. Patients who demonstrate at least minimal improvement after 12 weeks are randomly assigned to either continuing treatment at their current dose or switched to matching placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-65 years of age
* DSM-IV criteria for major depressive episode with atypical features as assessed by the Atypical Depression Diagnostic Scale
* minimum score of 18 on the Hamilton Depression Scale (29-item version) at baseline
* baseline Clinical Global Impressions Severity score of 4 or more
* written informed consent
* negative serum pregnancy test for women of childbearing potential

Exclusion Criteria:

* any current primary DSM-IV Axis I disorder other than depression
* history of DSM-IV diagnosis of bipolar I disorder, schizophrenia or other psychotic disorder, mental retardation or other pervasive developmental disorder, or cognitive disorder due to a general medical condition
* history of substance abuse or dependence within the last 3 months
* suicide risk or serious suicide attempt with the last year
* clinically significant medical condition or laboratory or EKG abnormality
* history of non-response to three prior adequate trials of antidepressants
* women of childbearing potential who are unwilling to practice an acceptable method of contraception
* history of hypersensitivity to modafinil
* use of an investigational medication within the last 28 days
* use of antidepressant medication with 28 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2003-02; Study Completion 2005-04

PRIMARY OUTCOMES:
HAM-D-29 (Hamilton Depression 29-Item Scale, with Atypical Features)

SECONDARY OUTCOMES:
ADDS (Atypical Depression Diagnostic Scale)
CGI-S (Clinical Global Impressions Severity Scale)
CGI-I (Clinical Global Impressions Improvement Scale)
SCL-90 (Symptom Checklist 90)
ESS (Epworth Sleepiness Scale)
BFI (Brief Fatigue Inventory)
FSS (Fatigue Severity Scale)
SOS (Severity of Symptoms Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, M.D., Principal Investigator — Duke Univeristy Medical Center